CLINICAL TRIAL: NCT05201131
Title: Canadian Cohort of Convective Thermal Therapy Using Rezūm System in Benign Prostatic Hyperplasia (BPH).
Status: Recruiting | Type: Observational
Sponsor: Can-Am HIFU Inc. (Other)
Responsible Party: Principal Investigator, Dean Elterman, Urologist, Can-Am HIFU Inc.
Other Study IDs: Rezum in BPH CAN
Record Dates: First submitted 2021-11-27; First posted 2022-01-21 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Urologic Diseases
Keywords: benigh prostate hypertrophy
MeSH Terms: conditions — Urologic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rezum procedure
  Interventions: Procedure: Rezum

INTERVENTIONS:
Procedure: Rezum — Rezum

SUMMARY:
To document the clinical outcome of Rezūm therapy for BPH patient in Canadian cohort.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects of ≥ 18 years of age.
* Primary diagnosis of Benign Prostate Hypertrophy (BPH).
* Candidate for Rezūm therapy as per clinical decision of Investigator.
* Willing and able to accurately complete the required questionnaires.
* Willing and able to provide signed and dated informed consent

Exclusion Criteria:

* Characteristics indicating a poor compliance with study protocol requirements.
* Disease or other health condition that is not suitable for this study.
* Unable or unwilling to provide signed informed consent.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — self-representation
Study Population: * Male subjects of ≥ 18 years of age.
  * Primary diagnosis of Benign Prostate Hypertrophy (BPH).
  * Candidate for or have already completed Rezūm therapy as per clinical decision of Investigator.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-10-07 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum flow rate (Q-max) | Baseline
  Maximum flow rate (Q-max)
Change of Maximum flow rate (Q-max) | 1 month after surgery
  Change of Maximum flow rate (Q-max)
Change of Maximum flow rate (Q-max) | 3 months after surgery
  Change of Maximum flow rate (Q-max)
Change of Maximum flow rate (Q-max) | 6 months after surgery
  Change of Maximum flow rate (Q-max)
Change of Maximum flow rate (Q-max) | 12 months after surgery
  Change of Maximum flow rate (Q-max)
Change of Maximum flow rate (Q-max) | 24 months after surgery
  Change of Maximum flow rate (Q-max)
Change of Maximum flow rate (Q-max) | 36 months after surgery
  Change of Maximum flow rate (Q-max)
Post-Void Residual (PVR) volume | Baseline
  Post-Void Residual (PVR) volume
Change of Post-Void Residual (PVR) volume | 1 month after surgery
  Change of Post-Void Residual (PVR) volume
Change of Post-Void Residual (PVR) volume | 3 months after surgery
  Change of Post-Void Residual (PVR) volume
Change of Post-Void Residual (PVR) volume | 6 months after surgery
  Change of Post-Void Residual (PVR) volume
Change of Post-Void Residual (PVR) volume | 12 months after surgery
  Change of Post-Void Residual (PVR) volume
Change of Post-Void Residual (PVR) volume | 24 months after surgery
  Change of Post-Void Residual (PVR) volume
Change of Post-Void Residual (PVR) volume | 36 months after surgery
  Change of Post-Void Residual (PVR) volume
Prostate Volume measured by transrectal ultrasound (TRUS) | Baseline
  Prostate Volume measured by transrectal ultrasound (TRUS)
Change of Prostate Volume measured by transrectal ultrasound (TRUS) | 12 months after surgery
  Change of Prostate Volume measured by transrectal ultrasound (TRUS)
Questionnaire | Baseline
  IPSS
Change of Questionnaire | 1 month after surgery
  Change of IPSS score
Change of Questionnaire | 3 months after surgery
  Change of IPSS score
Change of Questionnaire | 6 months after surgery
  Change of IPSS score
Change of Questionnaire | 12 months after surgery
  Change of IPSS score
Change of Questionnaire | 24 months after surgery
  Change of IPSS score
Change of Questionnaire | 36 months after surgery
  Change of IPSS score
Adverse Events | Baseline
  Adverse Events
Change of Adverse Events | 1 month after surgery
  Change of Adverse Events
Change of Adverse Events | 3 months after surgery
  Change of Adverse Events
Change of Adverse Events | 6 months after surgery
  Change of Adverse Events
Change of Adverse Events | 12 months after surgery
  Change of Adverse Events
Change of Adverse Events | 24 months after surgery
  Change of Adverse Events
Change of Adverse Events | 36 months after surgery
  Change of Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Dean Elterman, Principal Investigator — University Health Network, Toronto
Locations (1):
- Dean Elterman, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided